CLINICAL TRIAL: NCT06682767
Title: A Nutritional Intervention for Body, Brain, and Longevity Effects (NIBBLE) - A Randomized Open-label Intervention of the Fasting-mimicking Diet (FMD)
Brief Title: A Nutritional Intervention for Body, Brain, and Longevity Effects (NIBBLE)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Mitzi Gonzales, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00003359
Record Dates: First submitted 2024-10-29; First posted 2024-11-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cerebral Blood Flow; APOE 4
Keywords: APOE 4; prevention; nutritition; fasting mimicking diet; diet; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: As diet requires volitional activity, the study participants cannot be blinded. To minimize bias, the investigators evaluating cognitive, research labs, and MRI outcomes will be blinded to group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMD - Intervention (Experimental): Participants in the FMD group will be asked to refrain from consuming any calorie-containing foods or drinks other than the provided study foods/drinks during the designated intervention days each month.
  Interventions: Dietary Supplement: FMD1 (LNT22-017-1)
- Dietary Guidance (Active Comparator): The Dietary Guidance Group will receive nutrition recommendations based on the Harvard Healthy Eating Plate.
  Interventions: Behavioral: Dietary Guidance

INTERVENTIONS:
Dietary Supplement: FMD1 (LNT22-017-1) — FMD is a plant-based ketogenic diet that provides essential nutrients while maintaining hypo-caloric content. FMD is administered cyclically with 3-5 consecutive days of the diet followed by resumption of normal eating.
  Arms: FMD - Intervention
Behavioral: Dietary Guidance — Participants will receive established dietary guidance based on the Harvard Healthy Eating Plate.
  Arms: Dietary Guidance

SUMMARY:
The study aims to evaluate the safety, feasibility, and preliminary efficacy of six-month fasting-mimicking (FMD) relative to Dietary Guidance intervention in middle-aged adults at elevated risk for Alzheimer's disease due to the apolipoprotein (APOE) ε4 allele. Participants randomly assigned to the FMD intervention will consume a FMD for 5-days each month over a period of 6-months.

DETAILED DESCRIPTION:
Participants assigned to the FMD arm will adhere to the diet for 5 days a month over a period of 6-months. The FMD diet is produced by L-Nutra and provides 1100 kcals on the day 1 and 800 kcals on days 2-5. The diet consists of ingredients which are Generally Regarded As Safe (GRAS) selected for their fasting mimicking properties. The Dietary Guidance Group will receive recommendations based on the Harvard Healthy Eating Plate.

The overarching hypothesis of the study is that FMD relative to dietary guidance will be safe and well-tolerated. It is also hypothesized that FMD will be associated with increases in cerebral blood flow. . This is a phase 2 single-site trial with a randomized, open label, parallel assignment design. To minimize bias, individuals evaluating the cognitive, research lab, and MRI outcomes will be blinded to the assigned intervention group.

The study will enroll 40 participants who will be randomized 1:1 to the fasting-mimicking diet (FMD) intervention versus the Dietary Guidance group with stratification for age and sex. The intervention period is 6-months. Study visits 2-7 occur the day after the participant completes five days of FMD for that cycle if assigned to the FMD group. Visits 2, 3, 5, and 6 will be completed via phone or secure video platform. The intervention period is followed by a 3-month observational follow-up period for both groups.

The study design will enable preliminary investigations of the efficacy of FMD relative to the Dietary Guidance group for cognition, ADRD blood biomarkers, epigenetic clock, and brain structure in function in middle-aged adults at elevated risk for Alzheimer's disease due to the APOE e4 genotype. As diet requires volitional activity, the study participants cannot be blinded. To minimize bias, the investigators evaluating cognitive, research labs, and MRI outcomes will be blinded to group assignments.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 45-65 years at screening
4. Carrier of at least one copy of the APOE e4 allele
5. BMI 20-39kg/m2 (inclusive) at screening
6. On a stable medication regimen for at least 3 months.

Exclusion Criteria:

* Has any medical disease or condition that, in the opinion of the principal investigator (PI) or appropriate study personnel, precludes study participation* (*Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial);
* Significant depression (PHQ-9>9) or generalized anxiety (GAD-7>9)
* Diagnosis of a significant neurological condition such as multiple sclerosis, epilepsy, Parkinson's disease, major stroke
* Contraindications to MRI such as claustrophobia, cardiac pacemaker, etc.
* Current adherence or adherence within the past 3 months to a specialized diet (e.g. ketogenic, paleo, intermittent fasting, raw food, vegan)
* Food allergies (e.g. dairy, eggs, fish/shellfish, peanuts, tree nuts, soy, wheat, sesame, corn)
* Diagnosis of mild cognitive impairment or dementia; use of an FDA-approved medication for Alzheimer's disease; MoCA<23
* Diabetes (hbA1c >6.5%) or anti-diabetic medications
* History of gastric bypass;
* Inflammatory bowel disease
* Small or large bowel resection
* Subjects with recent weight loss (>5%), use of weight loss medication, participated in a weight loss program in the past 3 months
* Use of immune suppression drugs;
* Contraindication for study foods (special food needs and allergy);
* Women who are pregnant, lactating, or trying to conceive
* Alcohol dependency (alcohol intake greater than two drinks per day for women and three drinks per day for men)
* Current smoker or tobacco use within 3 months.
* Active malignant cancer or history of malignancy within the last 1 yea1s (except non-melanoma skin cancer)
* Serious psychiatric disorders such as schizophrenia, bipolar disorder, eating disorders
* Persons with allergy to animal dander or animal-instigated asthma

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of a six-month FMD intervention | From pre- to post-treatment (Day 165 +/-8 days)
  Endpoint: Number of adverse events in the intervention group relative to the Dietary Guidance group

SECONDARY OUTCOMES:
Investigate the impact of the FMD intervention on cerebral blood flow relative to the Dietary Guidance Group | From pre- to post-treatment (Day 165 +/-8 days)
  Endpoint: Cerebral blood flow - Cerebral blood flow will be assessed through brain magnetic resonance imaging arterial spin labeling sequence.
Investigate the impact of the FMD intervention on cognition relative to the Dietary Guidance group. | From pre- to post-treatment (Day 165 +/-8 days)
  NIH Toolbox Flanker and Pattern Comparison Tests and the Mayo Preclinical Alzheimer's Cognitive Composite.
  The NIH Toolbox assessments are measured through scaled scores (T-scores), which range from 20-80 with higher scores indicating better outcomes. The Mayo Preclinical Alzheimer's Cognitive Composite is also measured using a standardized score (Z-score) with mean of 0 and a standard deviation of 1. Higher scores indicate better performance.

OTHER OUTCOMES:
Examine the impact of FMD relative to Dietary Guidance on ADRD blood-based biomarkers | From pre- to post-treatment (Day 165 +/-8 days)
  Endpoint: Circulating levels of phosphorylated tau 217 (p-tau 217), neurofilament light (NFL), and glial fibrillary acidic protein (GFAP). The same unit of measurement applies for all - pg/ml.
Evaluate the efficacy of FMD relative to Dietary Guidance for modulating autophagic flux | From pre- to post-treatment (Day 165 +/-8 days)
  Endpoint: Autophagic flux in PBMCs and tissue (optional) Autophagy related gene expression. Both have the same unit of measurement as arbitrary units.
Evaluate the efficacy of FMD relative to Dietary Guidance for modulating insulin growth factor-1 | From pre- to post-treatment (Day 165 +/-8 days)
  Endpoint: insulin growth factor 1 (unit of measure is ng/ml)
Examine the impact of FMD relative to Dietary Guidance on systemic markers of inflammation through physiological parameters. | From pre- to post-treatment (Day 165 +/-8 days)
  Endpoint: Proteomic expression of pro-inflammatory markers Pro-inflammatory markers are IFN-γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, TNF-α, which are all measured in pg/ml.
Evaluate the efficacy of FMD relative to Dietary Guidance on epigenetic clock | From enrollment to end of study (Day 165 +/-8 days)
  Endpoint: Epigenetic modifications in peripheral blood mononuclear cells (unit of measure is DNA methylation age acceleration)
Evaluate the efficacy of FMD relative to Dietary Guidance for fasting blood glucose levels | From pre- to post-treatment (Day 165 +/-8 days)
  Endpoint: blood glucose (mg/dl)
Evaluate the efficacy of FMD relative to Dietary Guidance for body composition | From pre- to post-treatment (Day 165 +/-8 days)
  Endpoint: percent body fat and muscle mass (measure of unit: %)

CONTACTS AND LOCATIONS:
Overall Officials: Mitzi Gonzales, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be analyzed and stored at Cedars Sinai. After the study is completed, the de-identified, archived data will be stored at Cedars Sinai for use by other researchers including those outside of the study. As new relevant methodologies are developed, however, there is a conceivable future interest to process deidentified samples and data in a collaborating laboratory at Cedars-Sinai Medical Center or outside of Cedars-Sinai Medical Center including commercial entities. Participants are made aware of this possibility in the written informed consent form at the time of enrollment and are informed that to consent to this study is also to consent to permit coded data to be shared for the purposes of this research. The key to the code is not shared with collaborators but will remain in a HIPAA-compliant, secure, REDCap database at Cedars-Sinai Medical Center.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified data will be available within 6 months of release of the primary endpoint results and will be made available by request indefinitely
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and execution of a Data Sharing Agreement (DSA)